CLINICAL TRIAL: NCT05184985
Title: Efficacy of TrueRelief as a Non-Pharmacological Alternative for Pain Relief in Supraspinatus Tendonitis
Brief Title: TrueRelief Efficacy for Supraspinatus Tendonitis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was closed due to recruitment challenges. The study design involved frequent visits 3 times a week for 3 consecutive weeks which many prospective participants were not able to commit to.
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: TrueRelief, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21-01023230
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Supraspinatus Tendinitis; Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Intervention Model Description: Double blind, randomized, sham-controlled trial parallel arm study using TrueRelief as the experimental treatment and a TrueRelief device with sham capabilities as a placebo.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Placebo (Sham Comparator): Patients receive a placebo procedure using a sham TrueRelief device that looks and operates identically to the experimental TrueRelief device but will not emit any high frequency current.
  Interventions: Device: Sham TrueRelief device
- Experimental (Experimental): Patients receive an experimental procedure using a TrueRelief device.
  Interventions: Device: TrueRelief device

INTERVENTIONS:
Device: TrueRelief device — TrueRelief is an FDA-cleared treatment for chronic intractable pain, and as an adjunctive procedure in the management of post-surgical and post-traumatic acute pain. This 20,000 Hz high frequency electrical procedure is provided by clinicians trained in the use of the device and delivered via handheld steel-tipped probes to the source of pain and where pain is experienced.
  Arms: Experimental
Device: Sham TrueRelief device — The placebo device looks and operates identically to the experimental TrueRelief device but will not emit any high frequency current.
  Arms: Placebo

SUMMARY:
The investigators hypothesize that TrueRelief will result in improved outcomes for patients with shoulder pain compared to those receiving the sham TrueRelief treatment. Also, it is likely that those with fewer medical comorbidities will experience the greatest improvement.

DETAILED DESCRIPTION:
Supraspinatus tendonitis (SST) is a common source of shoulder pain that primary care, sports medicine, and orthopedic surgeons regularly manage. TrueRelief's FDA-cleared device, called TrueRelief 1250, is a noninvasive technology that provides pain relief through the delivery of high frequency pulsed direct electrical current to the skin surface around the location of the tendonitis via anode and cathode probes. This study will assess if TrueRelief may be an effective option in treating SST, given the preliminary data surrounding its anti-inflammatory and subsequent analgesic properties. The investigators are proposing the first double-blind, randomized, sham-controlled study of TrueRelief to determine a more accurate measurement of its efficacy, specifically in patients with SST. The investigators hypothesize that TrueRelief will result in improved outcomes in this patient population compared to those receiving the sham TrueRelief treatment.

ELIGIBILITY:
Inclusion Criteria:

* Those with shoulder pain of recent onset (<3 months)
* Those with supraspinatus tendonitis only (see exclusion criteria below)
* Those whose physical examination meets either criteria below:

  * Positive impingement tests
* At least two of:

  * Jobe
  * Modified Jobe
  * Hawkins-Kennedy
  * Neer
  * Painful arc:
* Painful arc at 70-120 degrees abduction and/or
* Painful arc at 70-120 degrees flexion
* Pain with resisted abduction and/or external rotation
* Those between the ages of 18 and 65
* Those willing and able to sign consent

Exclusion Criteria:

* Those who have had ipsilateral shoulder surgery involving the supraspinatus muscle
* Those who have experienced a fracture or avulsion fracture of any element of the shoulder or forequarter area (rib cage, clavicle, or humerus)
* Those with full-thickness rotator cuff tear
* Those with a long head of biceps rupture
* Those with shoulder pathology other than SST (ex: glenohumeral joint (GHJ) arthritis, adhesive capsulitis, labral tear). However, ACJ arthritis can be admitted since this is a very common comorbidity.
* Those with comorbidities that may confound the outcome, such as:

  * Diabetes (either type I or type II)
  * Auto-inflammatory diseases
  * Auto-immune diseases
  * Connective tissue disorders (Ehlers Danlos Syndrome)
* Those with demand type pacemakers
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change in pain measurements in patients with Supraspinatus Tendonitis (SST). | Beginning of study (Visit 1 - Week 1), Midpoint of Study (Visit 5 - Week 2), End of study (Visit 9 - Week 3), 1-month post-treatment follow-up call (Week 7-9)
  An assessment of the effect of TrueRelief on pain in patients with SST will be done by measuring pain at baseline, midpoint and at the end of the study treatment, as well as during the 1-month post-treatment follow-up phone call. Patients will be asked to rate their pain on a Visual Analog Pain Scale from 0 to 10, with 0 indicating no pain and 10 indicating emergency pain.

SECONDARY OUTCOMES:
Change in perceived shoulder function as measured by QuickDASH Questionnaire in patients with Supraspinatus Tendonitis (SST). | Beginning of study (Visit 1 - Week 1), Midpoint of Study (Visit 5 - Week 2), End of study (Visit 9 - Week 3), 1-month post-treatment follow-up call (Week 7-9)
  An assessment of the effect of TrueRelief on perceived function in patients with SST will be done through a QuickDASH questionnaire. This questionnaire will be administered at baseline, midpoint and at the end of the study treatment, as well as during the 1-month post-treatment follow-up phone call. The quickDASH questionnaire will be scored on a scale ranging from 0 (no disability) to 100 (most severe disability).
Change in perceived shoulder function as measured by a Shoulder Rating Questionnaire in patients with Supraspinatus Tendonitis (SST). | Beginning of study (Visit 1 - Week 1), Midpoint of Study (Visit 5 - Week 2), End of study (Visit 9 - Week 3), 1-month post-treatment follow-up call (Week 7-9)
  An assessment of the effect of TrueRelief on perceived function in patients with SST will be done through a Shoulder Rating questionnaire. This questionnaire will be administered at baseline, midpoint and at the end of the study treatment, as well as during the 1-month post-treatment follow-up phone call. A total weighted score will be calculated based on the answers to the Shoulder Rating Questionnaire, with values ranging from 0 (less severe condition of shoulder) to 100 (more severe condition of shoulder)

CONTACTS AND LOCATIONS:
Overall Officials: Vandana Sood, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian/Weill Cornell Medical Center Rehabilitation Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No